CLINICAL TRIAL: NCT06628245
Title: Validity and Reliability of Dubousset Functional Test in Lumbar Spinal Stenosis
Brief Title: The Dubousset Functional Test in Lumbar Spinal Stenosis
Status: Not yet recruiting | Type: Observational
Sponsor: Alanya Alaaddin Keykubat University (Other)
Responsible Party: Principal Investigator, Ayse Unal, Associate Professor, Alanya Alaaddin Keykubat University
Other Study IDs: 30.09.2024/DFT
Record Dates: First submitted 2024-10-03; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Lumbar Spinal Stenosis
Keywords: Lumbar Spinal Stenosis; Functional Status; Dubousset Functional Test; Reliability; Validity
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to investigate the validity and reliability of Dubousset Functional Test in the patients with lumbar spinal stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years, diagnosed with chronic pain (more than three months) due to lumbar spinal stenosis.

Exclusion Criteria:

* Those with fractures, pregnancy, a disease that would prevent physical exertion, those with a body mass index (BMI) of 40 kg/m2 and above, and those with major musculoskeletal or neurological disorders that cause gait disturbance will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sixty patients with lumbar spinal stenosis.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Dubousset Functional Test | 10 minutes
  The four test components included the Up and Walking Test (unassisted sit-to-stand from a chair, walk forward/backward 5 meters [no turn], then unassisted stand-to-sit), Steps Test (ascend three steps, turn, descend three steps), Down and Sitting Test (stand-to-ground, followed by ground-to-stand, with assistance as needed), and Dual-Tasking Test (walk 5 meters forwards and back while counting down from 50 by 2).